CLINICAL TRIAL: NCT01255462
Title: A Multicenter, Open Label, Single Ascending Dose Study to Assess the Safety, Tolerability, and Serum Pharmacokinetics of Intravitreal LFG316 in Patients With Advanced Age-related Macular Degeneration
Brief Title: Intravitreal LFG316 in Patients With Advanced Age-related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLFG316A2102
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Advanced Age-related Macular Degeneration
Keywords: AMD,; ARMD,; Age-related Macular Degeneration,; Eye Disease,; Wet AMD,; Neovascular AMD,; Choroidal Neovascular Membrane,; Choroidal Neovascularization,; Drusen,; Geographic Atrophy,; Complement,; C5,; Antibody
MeSH Terms: conditions — Macular Degeneration; Eye Diseases; Choroidal Neovascularization; Geographic Atrophy

ARMS (4):
- LFG316 0.15mg (Experimental)
  Interventions: Biological: LFG316
- LFG316 0.5mg (Experimental)
  Interventions: Biological: LFG316
- LFG316 1.5mg (Experimental)
  Interventions: Biological: LFG316
- LFG316 5mg (Experimental)
  Interventions: Biological: LFG316

INTERVENTIONS:
Biological: LFG316
  Arms: LFG316 0.15mg
Biological: LFG316
  Arms: LFG316 0.5mg
Biological: LFG316
  Arms: LFG316 1.5mg
Biological: LFG316
  Arms: LFG316 5mg

SUMMARY:
This study will assess the safety, tolerability, and serum pharmacokinetics of intravitreal LFG316 in patients with advanced age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Male or female AMD patients 55 to 90 years old, inclusive. In either eye, diagnosis of geographic atrophy or choroidal neovascularization due to AMD
* ETDRS best corrected visual acuity of 60 letters or worse in the study eye.

Exclusion Criteria:

* Retinal disease other than AMD in study eye which, in the investigator's opinion, may pose a safety risk or interfere with the study.
* Choroidal neovascularization due to a cause other than AMD.
* In the study eye, media opacity that interferes with fundus imaging or is likely to require surgery during the study period.
* Any of the following treatments to the study eye within 14 days prior to dosing: ranibizumab (Lucentis), bevacizumab (Avastin), pegaptanib (Macugen), or other VEGF inhibitor; OR likely requirement for one of the above treatments within 14 days of LFG316 administration.
* Any of the following within 30 days prior to dosing: photodynamic therapy treatment in the study eye; extrafoveal or juxtafoveal thermal laser photocoagulation in the study eye; systemic or topical (ophthalmic) steroid use in the study eye; bacterial keratitis in the study eye; OR intraocular surgery (including cataract surgery) in the fellow eye.
* Any of the following within 90 days prior to dosing: intraocular surgery (including cataract surgery) in the study eye; OR intravitreal or periocular corticosteroid injection in the study eye.
* Participation in another interventional clinical study, or use of any experimental treatment for AMD or any other investigational new drug within 12 weeks prior to the start of study treatment. Clinical trials solely involving over-the-counter vitamins, supplements, or diets will not exclude the patients from study participation.
* Any medical condition likely to interfere with the patient's participation in the study, or likely to cause serious adverse events during the study.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of single intravitreal doses of LFG316 in patients with advanced age-related macular degeneration. | Day 1 to Day 85 (starting from the day of intravitreal injection until the end of the study)

SECONDARY OUTCOMES:
To evaluate the serum pharmacokinetic profile of single intravitreal doses of LFG316 in patients with advanced age-related macular degeneration. | Day 1 to Day 85 (starting from the day of intravitreal injection until the end of the study)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- United States (8):
  - Retinal Consultants of Arizona,, Phoenix, Arizona
  - Retina-Vitreous Associates Medical Group,, Beverly Hills, California
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Opthalmic Consultants of Boston, Boston, Massachusetts
  - Charlotte Eye, Ear, Nose and Throat Associates, Charlotte, North Carolina
  - Texas Retina Associates, Dallas, Texas
  - Retina Consultants of Houston, Houston, Texas